CLINICAL TRIAL: NCT03743077
Title: Fitness and Health in Individuals With a Spinal Cord Injury: a Prospective Study
Brief Title: Health in Individuals With a Spinal Cord Injury: a Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Martha Sliwinski, Associate Professor of Rehabilitation and Regenerative Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAQ8226
Record Dates: First submitted 2018-11-13; First posted 2018-11-15 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Spinal Cord Injuries
Keywords: Exercise; Respiratory training
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individuals with spinal cord injury (Experimental): Volunteers will participate in the the spinal mobility fitness training program which includes exercise training with inspiratory muscle training.
  Interventions: Behavioral: Exercise training including inspiratory muscle training

INTERVENTIONS:
Behavioral: Exercise training including inspiratory muscle training — Volunteers will participate in the the spinal mobility fitness training program for a frequency of one to 3 times a week with pre and post tests including four objective measures of function (timed t-shirt test, timed transfer test, four direction reach test and trunk test of strength) and a pre and post subjective interview. In addition to the program consenting volunteers will perform inspiratory muscle training as a home program and submit weekly diaries tracking their training. The inspiratory muscle trainer by Respironics provides specific pressure for inspiratory muscle strength and endurance, regardless of how quickly or slowly patients breathe. It exercises respiratory muscles and improves breathing. It Improves muscle strength and is easy to use.

SUMMARY:
Individuals with a spinal cord injury need to exercise regularly to prevent the decline of health that results from a sedentary lifestyle. The purpose of this investigation is to examine the effects of a pre-existing exercise program and respiratory training on measures of health and quality of life in individuals who elect to participate in an existing 8-week supervised exercise program.

DETAILED DESCRIPTION:
The life expectancy of individuals with spinal cord injuries (SCI) has increased over the past decade. Yet, this population continues to present with an increased risk of a number of secondary health conditions, many of which occur sooner and at a higher rate than the normative population. As a program established to address this post-rehabilitative exercise participation necessity, it is determined that the Spinal Mobility fitness program, if found effective, can have vast positive effects in addressing aspects of health, function fitness, and overall quality of life for individuals with SCI. In addition to the need for exercise respiratory training is an important component of prevention of illness in individuals with a spinal cord injury. Genitourinary, skin disease and respiratory disorders are the top 3 reasons. Developing effective respiratory training programs in addition to exercise programs are critical for the prevention of illness and enabling a high quality of life. Pneumonia and septicemia are the two leading causes of decreased life expectancy in this population. Adding respiratory training to the spinal mobility program would be an appropriate intervention to further prevent health decline in these individuals.The spinal mobility course runs for eight weeks two times each year for 8 sessions for 4 to 5 hours each on Saturdays. Additionally individuals can participate in spinal mobility fitness training up to 3 times a week for one to three hours.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Individuals with spinal cord injury
* Medically stable
* Able to participate in the spinal mobility program

Exclusion Criteria:

* Individual with spinal cord injury who is medically unstable
* Cannot participate in an exercise program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-09-10 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Mean Time (seconds) for T-shirt Test | Up to 16 weeks post-intervention
  This test is designed to measure seated stability, and ability to maintain stability when performing an upper extremity task common in every day activities. At all times there are two researchers ready to assist subject should they lose their balance. Each subject is given two trials per testing period, and the average time is recorded. Shorter times indicate better performance.
Mean Time for Transfer Test | Up to 16 weeks post-intervention
  Subjects will execute transfer from and to the wheelchair in their normal fashion. They will be timed as they transferred to the mat table and from lying down back to the wheelchair. The time to perform these 2 tasks will be added as a single score. Each subject will perform 3 trials, and the mean time will be recorded.
Sitting Balance Performance Protocol, 4-way Reach Test | Up to 16 weeks post-intervention
  Measurements for excursion with an out stretched arm in the forward, backward and left and right lateral directions using a yard stick from start to maximal reach will be recorded.
Peak Force from Trunk Strength Test | Up to 16 weeks post-intervention
  Participants will instructed to sit in a posture that was as erect as possible. A hand held dynamometer (HHD) will be used to assess the strength. The HHD device will be placed between the examiner's hand and the participant's body with the force applied perpendicular to the trunk in four directions forward, backward, left and right. A second person will record the force values and guard the participant for safety purposes.

SECONDARY OUTCOMES:
Total Number of Respiratory Training Diaries Submitted | Up to 16 weeks post-intervention
  Compliance rate calculated by the total number of weekly sheets returned.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sliwinski, PT, PhD, MA, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center-NYPH, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Leathem JM, Macht-Sliwinski M, Boak S, Courville A, Dearwater M, Gazi S, Scott A. Community exercise for individuals with spinal cord injury with inspiratory muscle training: A pilot study. J Spinal Cord Med. 2021 Sep;44(5):711-719. doi: 10.1080/10790268.2019.1655200. Epub 2019 Sep 16. PMID 31525136